CLINICAL TRIAL: NCT02670954
Title: Evaluation of the Effect of Appropriate Sedation for Patients After Abdominal Surgeries : A Prospective Randomised Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Juanhong Shen, Director, PhD, Resident Physician, Principal Investigator, Chinese Medical Association
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Jinling37ICU
Record Dates: First submitted 2016-01-21; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Postoperative Sedation, Abdominal Surgery
MeSH Terms: interventions — Dexmedetomidine; Tramadol; Flurbiprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine,tramadol and flurbiprofen (Experimental): Both routine analgesic and sedation(dexmedetomidine,tramadol and flurbiprofen) are applied for this group of patients.
  Interventions: Drug: Dexmedetomidine, tramadol and flurbiprofen
- Tramadol and flurbiprofen (Active Comparator): Only routine analgesic(Tramadol and flurbiprofen) is applied for this group of patients.
  Interventions: Drug: tramadol and flurbiprofen

INTERVENTIONS:
Drug: Dexmedetomidine, tramadol and flurbiprofen
  Arms: Dexmedetomidine,tramadol and flurbiprofen
Drug: tramadol and flurbiprofen
  Arms: Tramadol and flurbiprofen

SUMMARY:
To evaluate the efficacy and safety of appropriate postoperative sedation with dexmedetomidine for patients after abdominal surgeries.Prospective randomised controlled study was conducted among patients after abdominal surgeries began in October 2015.The investigators enroll patients who received abdominal surgeries. One group receive sedative along with analgesic and the other group analgesic only for the other group on the first 24 hours after surgeries and will follow up for 3 days.

ELIGIBILITY:
Inclusion Criteria

* 16-85 years old
* underwent abdominal surgeries including enterectomy, gastrectomy, hepatectomy and pancreatectomy in the hospital and operation duration lasted at least 2 hours.

Exclusion Criteria

* take part in other clinical trials
* quinolone antibiotics intake 4 weeks prior to or within the study
* NSAIDS intake within one month
* history of peptic ulcer
* respiratory insufficiency
* renal insufficiency
* acute hepatitis or severe liver disease (Child-Pugh class C)
* pregnancy or lactation
* abnormal ECG with clinical significance
* uncontrolled hypotension
* bleeding tendency or hematological diseases
* untreated mechanical intestinal obstruction
* unable to express or any kind of mental disease.

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 1-3d after abdominal surgeries
  assessed by Prince Henry Pain Scale by investigators at 8:00 am after surgeries until discharge from ICU
recovery of gastrointestinal function | from admission to 30 days after abdominal surgeries
  assessed by time to first defecation
white blood cell count(10^9 /L) | 1-3d after abdominal surgeries
  evaluation of postoperative inflammatory response, blood sample collected at 6:00am for 1-3d after surgeries
C-reactive protein(mg/L) | 1-3d after abdominal surgeries
  evaluation of postoperative inflammatory response, blood sample collected at 6:00am for 1-3d after surgeries

SECONDARY OUTCOMES:
percentage of time within target sedation range | 1-3d after abdominal surgeries
  assessed by Richmond Agitation-Sedation Scale by investigators at 8:00 am after surgeries until discharge from ICU, target range is -2 to +1
risk of hypotension requiring interventions | 1-3d after abdominal surgeries
  systolic blood pressure <80 mmHg or/and diastolic blood pressure <50 mmHg is considered hypotension
risk of bradycardia requiring interventions | 1-3d after abdominal surgeries
  heart rate <40/min is considered bradycardia
use of opioids and use of benzodiazepins | 1-3d after abdominal surgeries

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of General Surgery of Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
basic characteristics of participant,interventions, primary and secondary outcomes, main results